CLINICAL TRIAL: NCT00002372
Title: A Phase I/II Screening Trial to Identify Potential Partner Compounds to Use in Combination With 141W94
Brief Title: A Study of 141W94 in Combination With Other Anti-HIV Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 264A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Administration, Oral; HIV Protease Inhibitors; Indinavir; Saquinavir; Nelfinavir; VX 478
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; amprenavir; Nelfinavir; Saquinavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Amprenavir
Drug: Nelfinavir mesylate
Drug: Saquinavir

SUMMARY:
To determine the steady-state pharmacokinetics of 141W94 in combination with saquinavir, indinavir and nelfinavir after multiple oral dosing. To determine the steady-state pharmacokinetics of saquinavir, indinavir, and nelfinavir in combination with 141W94 after multiple oral dosing. To assess the safety and tolerability of multiple doses of 141W94 when combined with saquinavir, indinavir and nelfinavir.

DETAILED DESCRIPTION:
Patients will be randomized to receive open label 141W94 in combination with saquinavir, indinavir and nelfinavir. The randomized phase will be preceded by a single dose pharmacokinetic interaction study of 141W94 and indinavir in 12 patients. Data from this single dose investigation will be used to determine the dose of indinavir to be used in the randomized phase.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed provided used with caution:

Medications that may interact at CYP3A4 (either a substrate, inhibitor or inducer of the enzyme) should be used with caution.

Patients must have:

* Documented HIV infection.
* CD4+ cell count >= 200 cells/mm3.

  1. Anticipated need for treatment with cytotoxic chemotherapeutic agents within the study time period.
* Treatment with immunomodulating agents.
* Medications that should not be administered with 141W94:

Terfenadine. Astemizole. Cisapride. Triazolam. Midazolam. Ergotamine/Dihydroergotamine-containing regimens. Antiretroviral drugs. Vitamin E supplements. Other experimental agents.

Anticipated need for radiation therapy within the study time period.

1. Prior protease inhibitors.

* Antiretroviral therapy within 2 weeks prior to entry.
* Treatment with cytotoxic chemotherapeutic agents within 4 weeks prior to entry.

Radiation therapy within 4 weeks prior to entry. Current alcohol or illicit drug use that, in the opinion of the investigator, may interfere with the patient's ability to comply with the dosing and protocol evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - ViRx Inc, San Francisco, California
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] Eron JJ, Haubrich R, Lang W, Pagano G, Millard J, Wolfram J, Snowden W, Pedneault L, Tisdale M. A phase II trial of dual protease inhibitor therapy: amprenavir in combination with indinavir, nelfinavir, or saquinavir. J Acquir Immune Defic Syndr. 2001 Apr 15;26(5):458-61. doi: 10.1097/00126334-200104150-00008. PMID 11391165